CLINICAL TRIAL: NCT01444235
Title: A Prospective Randomized Double Blind Multicenter Phase III Study Comparing Two Methods of Cardioplegia in Coronary Artery Bypass Surgery Custodiol-N Versus Custodiol
Brief Title: Phase III Study Comparing Two Methods of Cardioplegia in Coronary Artery Bypass Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. F. Köhler Chemie GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-N-CSM-III/01/08
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: CAD, ACVB
MeSH Terms: conditions — Coronary Artery Disease | interventions — Custodiol-N solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Custodiol (Active Comparator): After cross clamping of the aorta on cardiopulmonary bypass, the Custodiol solution, at a temperature of 4 - 6°C, will be infused antegrade into the root of the aorta.
  Interventions: Drug: Custodiol
- Custodiol-N (Experimental): After cross clamping of the aorta on cardiopulmonary bypass, the Custodiol-N solution, at a temperature of 4 - 6°C, will be infused antegrade into the root of the aorta.
  Interventions: Drug: Custodiol-N

INTERVENTIONS:
Drug: Custodiol-N — Route of administration: by infusion Dosage: will be infused antegrade into the root of the aorta until 1500-2000 mL of solution have been infused Duration: infusion technique will be continued for seven minutes
  Arms: Custodiol-N
Drug: Custodiol — Route of administration: by infusion duration: infusion technique will be continued for seven minutes dosage: until 1500-2000 mL of solution have been infused
  Arms: Custodiol

SUMMARY:
Comparison of the cardioprotective effects and safety of two cardioplegic solutions (solutions used during a cardiac arrest in the heart surgery) in patients undergoing cardiopulmonary bypass for coronary artery bypass surgery.

DETAILED DESCRIPTION:
The objective of this investigation is to compare the cardioprotective effects and safety of two cardioplegic solutions, HTK Cardioplegic Solution (Custodiol) and Custodiol-N in patients undergoing cardiopulmonary bypass for coronary artery bypass surgery. The study design is a prospective, double blind, multicenter, randomized, Phase III comparison study intended to demonstrate non-inferiority in surgical outcome between Custodiol and Custodiol-N as determined by CK-MB area under the curve (primary endpoint), catecholamine requirement(cumulative dose) and cardiac Troponin T, occurrence of comorbid events postoperatively (e.g., myocardial infarction).

ELIGIBILITY:
Inclusion Criteria:

The study population will be selected from patients of either sex with coronary artery disease (CAD) who are to undergo cardiopulmonary bypass for coronary artery bypass surgery.

1. Patients >/=35 and </=80 years of age
2. Male or female with 2 or 3 vessel coronary disease, who are scheduled for elective CBP surgery for coronary revascularisation
3. Presence of definite CAD for which surgical intervention is deemed necessary, without evidence of ongoing infarction.

   Patients with unstable angina can be included as long as there is no objective (negative cardiac isoenzymes in the immediate six hours preceding CABG, current intravenous use of nitrate therapy) or subjective (absence of prolonged symptoms suggestive of coronary insufficiency that do not respond to pharmacologic intervention) evidence of myocardial necrosis.
4. Eligibility for Swan-Ganz-Catheter
5. Able to understand character and individual consequences of the clinical trial and to provide written informed consent to participate in the study
6. No evidence of severe organic or psychiatric disease by history or physical examination
7. No history of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or no any history of drug abuse or addiction within 12 months of study enrollment.

Exclusion Criteria:

1. Patients undergoing valve repair or replacement
2. History of recent (< 6 weeks) Q-wave myocardial infarction
3. Left ventricular ejection fraction < 35% (as assessed by any one of the following: contrast ventriculography, multigated acquisition scanning [MUGA], or 2-D ECHO)
4. Patients on intra-aortic balloon devices or with history of previous coronary artery bypass surgery
5. Pregnant or lactating patients
6. Patients who have participated in any other investigational studies within 30 days previous to enrollment
7. Patients in cardiogenic shock (defined as a systolic BP < 90 mmHg for over one hour despite inotropic and chronotropic support)
8. Patients with severe chronic obstructive lung disease (FEV1 < 50%)
9. Previous cardiac valvular disease (clinical relevant)
10. Dialysis or creatinine > 2 mmol/L
11. BMS-Stent < 4 weeks
12. DES-Stent < 6 month
13. Guidance depended Plavix therapy

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
CK-MB area under the curve within 24 hours | Up to 24 hours after the aortic clamp release
  Measurements will be carried out at the following timepoints: 4,8,12,16,20,24 hours (± 30 min) after release of the aortic cross clamp

SECONDARY OUTCOMES:
Catecholamine requirement | 24 hours (cumulative dose)
  Catecholamine requirement on surgical ICU within 24 hours
CK-MB peak | Up to day 5
  CK-MB peak on the days 2, 3, 4 and 5 after removal of aortic cross clamp
Mortality any time during post-op through Day 30 | Up to Day 30
  Mortality will be documented at any time during post-op through Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Szabo, Prof. Dr., Principal Investigator — Department of Cardiac Surgery of University of Heidelberg; Nikolaus Pizanis, Dr., Principal Investigator — Klinik für Thorax- und Kardiovaskuläre Chirurgie, Universitätsklinikum Essen; Florian Wagner, Dr., Principal Investigator — Klinik für Herz- und Gefäßchirurgie, Universitäts-Krankenhaus Eppendorf; Thorsten Doenst, Prof. Dr., Principal Investigator — Klinik für Herz- und Thoraxchirurgie, Universitätsklinikum Jena; Martin Misfeld, Dr., Principal Investigator — Herzzentrum Leipzig GmbH, Klinik für Herzchirurgie
Locations (4):
- Germany (4):
  - Klinik für Thorax- und Kardiovaskuläre Chirurgie, Universitätsklinikum Essen, Essen
  - Abt. Herzchirugie, Universitätsklinikum Heidelberg, Heidelberg
  - Klinik für Herz- und Thoraxchirurgie, Universitätsklinikum Jena, Jena
  - Herzzentrum Leipzig GmbH, Leipzig